CLINICAL TRIAL: NCT06619561
Title: A Phase 2, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, PK, and Efficacy of Vimseltinib in Adults With Active Chronic GVHD After Failure of Prior Systemic Therapy
Brief Title: A Study to Evaluate Vimseltinib in Adults With Active Chronic Graft-Versus-Host Disease (cGVHD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCC-3014-02-001
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Graft-Versus-Host Disease (cGVHD)
Keywords: Allogeneic hematopoietic stem cell transplant (HSCT); Graft-Versus-Host Disease; GVHD; cGVHD; Graft versus host disease; Immune System Diseases; Organizing Pneumonia; Bronchiolitis Obliterans; Bronchiolitis; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Bronchiolitis Obliterans Syndrome; Graft vs Host Disease; Sclerosis; Fibrosis; Hematopoietic stem cell transplantation; Liver diseases
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Graft vs Host Disease; Immune System Diseases; Organizing Pneumonia; Bronchiolitis Obliterans; Bronchiolitis; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Sclerosis; Fibrosis; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vimseltinib (Experimental): Escalating doses of vimseltinib in 28 day cycles.
  Interventions: Drug: Vimseltinib

INTERVENTIONS:
Drug: Vimseltinib — Administered orally
  Other Names: DCC-3014

SUMMARY:
The purpose of this study is to determine if vimseltinib is safe, tolerable and works effectively to treat adults with active moderate to severe cGVHD. Participants will be treated with vimseltinib in 28-day treatment cycles for approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Must be allogeneic hematopoietic stem cell transplant (HSCT) recipients with moderate to severe cGVHD requiring systemic immune suppression.

   a. May have persistent active acute GVHD (aGVHD) and chronic GVHD (cGVHD) manifestations (overlap syndrome).
2. Participants with active cGVHD who have received and failed at least 2 prior lines of systemic therapy.
3. Stable dose of systemic corticosteroids is permitted but not required. If being taken, participants should be on a stable dose of corticosteroids for at least 2 weeks prior to starting study drug treatment.
4. Adequate organ and bone marrow functions.
5. Participants of reproductive potential agree to follow the contraception requirements.
6. Karnofsky Performance Scale (KPS) of ≥60.

Exclusion Criteria:

1. Has aGVHD without manifestations of cGVHD.
2. Prior use of colony-stimulating factor 1 receptor (CSF1R) inhibitor for cGVHD.
3. History or other evidence of severe illness, uncontrolled infection, or any other conditions that would make the participant unsuitable for the study. All wounds must be healed and free of infection or dehiscence.
4. History of malignancy except for:

   1. Underlying malignancy for which the transplant was performed
   2. Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to enrollment and felt to be at low risk for recurrence.
5. Malabsorption syndrome or other illness that could affect oral absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLTs) | Cycle 1 (28 Days)
  DLTs assessed for each dose level.
Number of Participants with Adverse Event(s) (AEs) and Serious Adverse Event(s) (SAEs) | Baseline to Study Completion (Estimated up to 24 months)
  AEs and SAEs assessed for each dose level.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline up to Cycle 7 Day 1 (Cycle = 28 days)
  ORR is percentage of participants achieving best overall response of complete response (CR) or partial response (PR) up to Cycle 7 Day 1 based on 2014 National Institutes of Health (NIH) cGVHD Criteria.
Duration of Response (DOR) | First CR or PR until PD or Death due to Any Cause (Estimated up to 24 months)
  DOR for participants with CR or PR, defined as the time interval from the time of first CR or PR per 2014 NIH cGVHD Criteria, until PD, initiation of new systemic therapy for cGVHD, or death due to any cause, whichever occurs first.
Organ-Specific Response | Baseline up to Cycle 7 Day 1 (Cycle = 28 days)
  Organ-specific response per 2014 NIH cGVHD Criteria up to Cycle 7 Day 1
Failure-Free Survival (FFS) | Baseline to, whichever occurs first of, PD, Addition of Systemic Immune Suppressive Therapy, or Death due to Any Cause (Estimated up to 24 months)
  FFS is the time from first dose to progressive disease (PD) per 2014 NIH cGVHD Criteria, initiation of new systemic therapy for cGVHD, or death due to any cause, whichever occurs first.
Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) | Estimated up to 24 months
  Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (26):
- United States (26):
  - City of Hope National Medical Center, Duarte, California
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - University of California Irvine Health, Orange, California
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Illinois Medical Center - Hematology & Oncology, Chicago, Illinois
  - University of Kansas Cancer Center-Westwood, Westwood, Kansas
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tristar Bone Marrow Transplant, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Intermountain Health, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia